CLINICAL TRIAL: NCT03416153
Title: A Multi-Center Phase II Trial of Individualized Adaptive De-escalated Radiotherapy Using Pre and Mid-Treatment FDG-PET/CT for HPV-related Oropharynx Cancer
Brief Title: Individualized Adaptive De-escalated Radiotherapy for HPV-related Oropharynx Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: VA Ann Arbor Healthcare System (U.S. Federal Agency); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2017.113; HUM00136258 (Other: University of Michigan); U01CA183848 (NIH)
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Results first posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Oropharynx Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Carboplatin; Radiotherapy; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Standard Treatment (Active Comparator): Patients will receive a single prescription of 70 Gy in 35 fractions with RT given once daily, 5 days a week along with weekly carboplatin and paclitaxel (standard therapy)
  Interventions: Drug: Carboplatin; Radiation: Radiation Therapy; Drug: Paclitaxel
- De-escalation Treatment (Experimental): Patients will initially receive a single prescription of 70 Gy in 35 fractions with RT given once daily, 5 days a week along with weekly carboplatin and paclitaxel (standard therapy). If certain parameters are met radiation therapy will be reduced to 54Gy to high risk Planned Target Volume (PTV) and 43.2Gy to low risk PTV all in 27 fractions.
  Interventions: Drug: Carboplatin; Radiation: Radiation Therapy; Drug: Paclitaxel

INTERVENTIONS:
Drug: Carboplatin — AUC=1 weekly during radiation therapy. Carboplatin will be given once a week in combination with paclitaxel (standard treatment), concurrent with radiation therapy. Given IV.
Radiation: Radiation Therapy — Patients will initially receive a single prescription of 70 Gy to PTV1 in 35 fractions with RT given once daily, 5 days a week along with weekly carboplatin and paclitaxel (standard therapy). Dose will be reduced to 54Gy to high risk PTV and 43.2Gy to low risk PTV all in 27 fractions for patients who meet pPET-CT and iPET-CT parameters.
Drug: Paclitaxel — 30 mg/m2 weekly during radiation therapy. Paclitaxel will be given once a week in combination with carboplatin (standard treatment), concurrent with radiation therapy. Given IV.

SUMMARY:
This prospective study aims to utilize pre- and mid-treatment PET-CT to guide de-escalation of radiation therapy in HPV-related squamous cell carcinoma of the oropharynx.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have FDG-avid and histologically or cytologically proven squamous cell carcinoma of the oropharynx (tonsil, base of tongue, oropharyngeal wall, soft palate) that is p16 positive by immunohistochemistry or HPV positive by in situ hybridization.
* AJCC eighth edition staging stage 1 and stage 2
* Appropriate stage for protocol entry, including no distant metastases, based upon the following minimum diagnostic workup:
* History/physical examination, including documentation of weight within 4 weeks prior to registration;
* FDG-PET/CT scan for staging and RT plan within 4 weeks prior to registration;
* Zubrod Performance Status (A quantification of the functional status of cancer patients that runs from 0 to 5, with 0 denoting perfect health and 5 death) 0-1 within 4 weeks prior to registration;
* Age ≥ 18;
* Able to tolerate PET/CT imaging required to be performed
* CBC/differential obtained within 4 weeks prior to registration on study, with adequate bone marrow function;
* Serum creatinine within normal institutional limits or a creatinine clearance ≥ 45 ml/min within 4 weeks prior to registration;
* Women of childbearing potential and male participants must agree to use a medically effective means of birth control throughout their participation in the treatment phase of the study.
* The patient must provide study-specific informed consent prior to study entry.

Exclusion Criteria:

* cT4, cN3 or cM1 disease
* "Matted nodes" as determined by review with Neuroradiology
* Gross total excision of both primary and nodal disease with curative intent; this includes tonsillectomy, local excision of primary site, and nodal excision that removes all clinically and radiographically evident disease. In other words, to participate in this protocol, the patient must have clinically or radiographically evident gross disease for which disease response can be assessed.
* Carcinoma of the neck of unknown primary site origin (even if p16 positive);
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years
* Any prior therapy for the study cancer; note that prior chemotherapy for a different cancer is allowable if > 3 years prior to study;
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields;
* Severe, active co-morbidity;
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception;
* Poorly controlled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2025-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Mierzwa, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (2):
- United States (2):
  - University of Michigan Hospital, Ann Arbor, Michigan
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 subjects were removed from the trial before being assigned a cohort.
Groups:
- Standard Treatment: Patients received a single prescription of 70 Gy in 35 fractions with RT given once daily, 5 days a week along with weekly carboplatin and paclitaxel (standard therapy)
  Carboplatin: AUC=1 weekly during radiation therapy. Carboplatin will be given once a week in combination with paclitaxel (standard treatment), concurrent with radiation therapy. Given IV.
  Radiation Therapy: Patients will initially receive a single prescription of 70 Gy to PTV1 in 35 fractions with RT given once daily, 5 days a week along with weekly carboplatin and paclitaxel (standard therapy). Dose will be reduced to 54Gy to high risk PTV and 43.2Gy to low risk PTV all in 27 fractions for patients who meet pPET-CT and iPET-CT parameters.
  Paclitaxel: 30 mg/m2 weekly during radiation therapy. Paclitaxel will be given once a week in combination with carboplatin (standard treatment), concurrent with radiation therapy. Given IV.
- De-escalation Treatment: Patients initially received a single prescription of 70 Gy in 35 fractions with RT given once daily, 5 days a week along with weekly carboplatin and paclitaxel (standard therapy). If certain parameters are met radiation therapy will be reduced to 54Gy to high risk Planned Target Volume (PTV) and 43.2Gy to low risk PTV all in 27 fractions.
  Carboplatin: AUC=1 weekly during radiation therapy. Carboplatin will be given once a week in combination with paclitaxel (standard treatment), concurrent with radiation therapy. Given IV.
  Radiation Therapy: Patients will initially receive a single prescription of 70 Gy to PTV1 in 35 fractions with RT given once daily, 5 days a week along with weekly carboplatin and paclitaxel (standard therapy). Dose will be reduced to 54Gy to high risk PTV and 43.2Gy to low risk PTV all in 27 fractions for patients who meet pPET-CT and iPET-CT parameters.
  Paclitaxel: 30 mg/m2 weekly during radiation therapy. Paclitaxel will be given once a week in combination with carboplatin (standard treatment), concurrent with radiation therapy. Given IV.
Period: Overall Study
Arm/Group | Standard Treatment | De-escalation Treatment
Started | 49 | 36
Completed | 47 | 35
Not Completed | 2 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment | De-escalation Treatment | Total
Number analyzed (Participants) | 49 | 36 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 23 | 54
  >=65 years | 18 | 13 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 43 | 34 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 47 | 36 | 83
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 47 | 33 | 80
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 49 | 36 | 85

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients With Local Regional Recurrence (LRR) of Disease
Description: RECIST (Response Evaluation Criteria In Solid Tumors) will be used to evaluate response and recurrence. All patients will be analyzed together as the goal of the study is to estimate risk of LRR in this patient population treated with this particular strategy in which some patients continue to receive standard therapy while others are de-escalated. Results will also be estimated and reported separately for patients receiving standard or de-escalated therapy.
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standard Treatment | De-escalation Treatment
Number analyzed (Participants) | 49 | 36
percentage of participants | 2 [0 to 6] | 3 [0 to 8]

2. Primary Outcome: Change in Metabolic Tumor Volume 50% (MTV 50%)
Description: The change in metabolic tumor volume (MTV)50% at the mid-treatment timepoint will be calculated as percent change from baseline and used as a continuous variable in a Cox model for an outcome of time to LRR. Will also evaluate more non-parametrically, the relation between hazard of LRR and mid-treatment MTV50% using a kernel estimator in a Cox model.
Time Frame: 2 months
Population: 2 patients were not evaluable
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Standard Treatment | De-escalation Treatment
Number analyzed (Participants) | 47 | 36
percent change from baseline | -11.3 (66.7) | -71.1 (16.7)

3. Secondary Outcome: Quality of Life Assessed Per the Functional Assessment of Cancer Therapy-Head and Neck (FACTHN)
Description: Quality of life (QOL) outcomes and swallowing study results will be summarized descriptively by timepoint. If there is substantial missingness in the QOL outcomes the study will assess for informative missingness by comparing earlier QOL scores and change in earlier QOL scores between patients missing QOL at later time points (e.g. 1 or 2 years).
Time Frame: 2 Years
Reporting Status: Not Posted

4. Secondary Outcome: The Proportion of Patients Alive
Time Frame: 2 Years
Reporting Status: Not Posted

5. Secondary Outcome: Incidence of Toxicity
Description: Toxicity outcomes will be estimated as proportions of patients with available toxicity data at 3, 6 12 and 24 months.
Time Frame: 3, 6, 12 and 24 Months
Reporting Status: Not Posted

6. Secondary Outcome: Detectable Circulating Tumor Deoxyribonucleic Acid (ctDNA) in Participants
Description: The proportion of patients in whom ctDNA is detectable will be summarized as a binomial proportion at each timepoint. Additionally, the relation between ctDNA presence or other characteristics and patient outcomes including time to local or distant progression will be assessed by including ctDNA as a covariate in Cox models for local or distant control.
Time Frame: 4 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events and All-Cause Mortality have been reported through the time of PCC. Data is still being collected. Results currently reported were collected over a 5 year period.
Description: Adverse Events and All-Cause Mortality have been reported through the time of PCC. Data is still being collected.
Arm/Group | Standard Treatment | De-escalation Treatment
All-Cause Mortality (participants affected / at risk) | 2/49 | 1/36
Serious Adverse Events (participants affected / at risk) | 5/49 | 3/36
Other Adverse Events (participants affected / at risk) | 49/49 | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Treatment (N=49) | De-escalation Treatment (N=36)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Oral hemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Oral pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Treatment (N=49) | De-escalation Treatment (N=36)
Abdominal pain (General disorders) | 4 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (5) | 0 (0)
Anemia (Investigations) | 4 (5) | 0 (0)
Anorexia (Psychiatric disorders) | 7 (7) | 0 (0)
Anxiety (Psychiatric disorders) | 8 (8) | 0 (0)
Constipation (Gastrointestinal disorders) | 31 (38) | 18 (20)
Dehydration (General disorders) | 21 (27) | 6 (6)
Dermatitis radiation (Skin and subcutaneous tissue disorders) | 39 (75) | 25 (32)
Diarrhea (Gastrointestinal disorders) | 5 (7) | 7 (7)
Dizziness (General disorders) | 5 (5) | 4 (5)
Dry mouth (General disorders) | 46 (73) | 31 (45)
Dysgeusia (General disorders) | 49 (81) | 33 (51)
Dysphagia (General disorders) | 37 (66) | 24 (34)
Ear pain (Ear and labyrinth disorders) | 11 (12) | 8 (9)
Esophageal pain (Gastrointestinal disorders) | 27 (35) | 5 (5)
Esophagitis (Gastrointestinal disorders) | 4 (4) | 0 (0)
Fatigue (General disorders) | 48 (57) | 25 (31)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 0 (0)
Headache (General disorders) | 8 (9) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (6) | 0 (0)
Lymphedema (Vascular disorders) | 8 (8) | 0 (0)
Lymphocyte count decreased (Investigations) | 6 (17) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 45 (85) | 30 (39)
Nausea (Gastrointestinal disorders) | 32 (49) | 20 (23)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Oral pain (Musculoskeletal and connective tissue disorders) | 47 (80) | 25 (33)
Pain (General disorders) | 32 (59) | 26 (35)
Radiation recall reaction (dermatologic) (Skin and subcutaneous tissue disorders) | 4 (6) | 0 (0)
Sore throat (General disorders) | 19 (22) | 10 (10)
Thrush (Infections and infestations) | 7 (7) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 9 (10) | 4 (4)
Vomiting (Gastrointestinal disorders) | 4 (4) | 4 (5)
Weight loss (Investigations) | 36 (45) | 19 (20)
Hypotension (Vascular disorders) | 0 (0) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT03416153/Prot_SAP_001.pdf
  • Informed Consent Form (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT03416153/ICF_000.pdf